CLINICAL TRIAL: NCT04043884
Title: sEmg Biofeedback Training in Individuals With Subacromial Pain Syndrome: Randomized Controlled Trial
Brief Title: sEmg Biofeedback Training in Individuals With Subacromial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physical Therapy and Lab Head, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKAO2019
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Shoulder Pain
Keywords: Shoulder rehabilitation; Electromyography; Posture analysis
MeSH Terms: conditions — Shoulder Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sEmg Biofeedback training (Experimental): 8-week exercise program, twice a week, with emg biofeedback training.
  Interventions: Other: sEmg biofeedback training
- Exercises (Active Comparator): 8-week exercise program, twice a week.
  Interventions: Other: Strength training

INTERVENTIONS:
Other: sEmg biofeedback training — Volunteers will perform scapular strengthening and stabilization exercises added to sEMG biofeedback in the upper trapezius (TS), Trapezius (TM), Lower Trapezius (TI), and Serratil Anterior (AS) muscles in real time displayed in a Computer screen.
  Arms: sEmg Biofeedback training
Other: Strength training — The volunteers will perform a strengthening protocol with elbow flexion exercises, medial and lateral shoulder rotation, scapular retraction and push up plus.
  Arms: Exercises

SUMMARY:
Objective: To investigate the effects of EMG biofeedback training on the pattern of scapular muscle activation and kinematics in subjects with subacromial pain syndrome. Methods: This is a randomized controlled trial, which will be composed of 40 volunteers of both genders, aged between 30 and 60 years. All volunteers will undergo pre-assessment (IA): pain sensation, pain and function, shoulder range of motion, muscle strength, electromyographic activity and kinematics of the shoulder complex. After the initial evaluation, the volunteers will be randomly divided into two groups for the intervention: exercises group (GE - conventional exercises with elastic band) and Biofeedback group (BG - Biofeedback training). The intervention protocol will last eight weeks. After four weeks, the second assessment (SA), similar to IA, will be performed and the global change perception questionnaire will be added. At the end of the intervention protocol, the third evaluation (TA), similar to SA, will be performed. A follow-up will be performed 4 weeks after the end of the intervention protocol, with the assessment being equal to TA. Statistical Analysis will be performed through Statistical Package for Social Sciences (SPSS) software version 20.0 for Windows, following the principles of intention-to-treat analysis. The descriptive analysis will use the mean as a measure of central tendency and the standard deviation as a measure of dispersion. A mixed model ANOVA will be performed for intra and intergroup comparisons.

DETAILED DESCRIPTION:
This work was submitted to the Ethics and Research Committee (CEP) of the Federal University of Rio Grande do Norte through the national interface "Plataforma Brasil" and approved in its ethical aspects based on Resolution 466/12 of the National Health Council and the Declaration of Helsinki under registration number 3246854. All data will be registered in a confidential database of the laboratory and can only be handled by the responsible researchers. All individuals will be invited to voluntarily participate in the study and must sign the Free and Informed Consent Form (FICF) containing information about the purposes, risks and benefits of the research. A pilot study was carried out aiming at the adequacy of all the research procedures, as well as the training of the researchers involved. After signing the FICF sociodemographic, anthropometric and clinical data will be collected and then the individuals will be submitted to the evaluation procedures. Four identical evaluations will be carried out before, during and after the intervention protocol. Initially, initial assessment (IA) will record the baseline data prior to the protocol, the second assessment (SA) will be performed after the first four weeks of protocol, the third (TA) at the end of the 8 week intervention protocol, and the fourth (FA) four weeks after the end of the protocol. The evaluation of the pain sensation will be performed through the numerical pain scale. Volunteers will be instructed by the evaluator to scale the intensity of pain based on the last 24 hours. The scale is composed of 11 items, 0 being described as "painless" and 10 as "worst possible pain" at its extremities. Participants will then complete the Brazilian version of the Desabilities of the arm, shoulder and Hand (DASH) questionnaire. It is a self-assessment questionnaire containing 30 questions with the purpose of assessing physical function, symptoms and social function. Five possible responses are presented ranging from "no difficulty" to "unable to perform activity". Responses are scored on a rating scale of one to five points. The score calculation is performed by applying established formulas. Volunteers will be instructed by the evaluator to complete the items in the questionnaire that have been applicable in the last 24 hours. The higher the final score, the greater the disability. Motion amplitudes will be evaluated by the Smartphone clinometer application (Plaincode Software Solutions) which operates as a reliable and validated inclinometer. The Range Of Motion (ROM) of flexion, hyperextension, lateral rotation and medial rotation of the shoulder will be evaluated. The flexion and the hyperextension of the shoulder will be evaluated in the sitting position. The evaluator will position the smartphone parallel to the subject's arm secured in an appropriate device, aligned to the lateral epicondyle of the elbow and will request flexion and active hyperextension respectively of the shoulder with the elbow in complete extension. Lateral and medial rotation of the shoulder will be evaluated with the volunteer in the supine position at the table, shoulder abducted at 90 ° and elbows at 90 ° flexion. The evaluator will position the smartphone on the forearm of the individual aligned between the lateral epicondyle and the wrist and between the medial epicondyle and the wrist for the medial and lateral rotation movement respectively. Peak torque evaluation will be perfomed using a portable hand held dynamometer (Lafayette Instrument®, model 01165, USA). Data will be recorded from two 5 seconds maximum voluntary isometric contractions (MVIC), with a 1-minute interval. The average of the two tests will be considered for analysis. The evaluation will be carried out by the same evaluator and will be positioned in such a way as to counteract the requested movement. The electromyographic signal will be captured by an 8-channel signal conditioning modulator (Noraxon® surface, Scottsdale, AZ, USA) with a 16-bit resolution and common mode rejection rate> 100 Db. The signals will be captured at a sample rate set to 1500 Hz, filtered at a frequency between 10 and 500 Hz and amplified 1000 times. Signal capture will be performed using passive surface self-adhesive electrodes (Noraxon®, USA), separated by an inter-electrode distance of 2 cm. The electrodes were placed in the Upper Trapezius (UT), Lower Trapezius (LT), Middle Trapezius (MT) and Serratus Anterior (SA) muscles, in accordance with the SENIAM guidelines . First, individuals will perform three movements of arm elevations in the plane of the scapula in the standing position. The arm will be positioned at 40 degrees from the frontal plane measured by MotionMonitor software (Innovative Sports Training, Chicago, IL) of kinematic analysis and the motion will be directed with the aid of a vertical support. Each movement should occur in approximately eight seconds with four seconds in the concentric phase and four seconds in the eccentric phase. The subjects will then perform isometric contractions of 5 seconds with and without load at angles 30 °, 60 °, 90 ° and 120 ° of shoulder abduction. The load will be determined from a test with the same movement with dumbbells of 2kg, 1kg and 0.5kg respectively Taking as reference a score not higher than 3 on the Borg effort scale (moderate effort). The Root Means Square averages for each phase will be recorded and the ratios UT / LT, UT / MT, UT / SA will be analyzed. The electromyographic data (in microvolts) will be normalized by the peak of the signal recorded during the MVIC. The three-dimensional analysis of the movement of the shoulder complex will be performed using the Flock of Birds (Ascension Technologies, Burlington, VT) electromagnetic tracking system associated with MotionMonitor software (Innovative Sports Training, Chicago, IL). Volunteers will be asked to stay in a neutral position with the transmitter directly in the shoulder joint to be evaluated and three superficial electromagnetic sensors will be positioned to the skin of the volunteers in pre-established anatomical marks. A double-sided tape will be used, in specific anatomical points: in the sternum, inferiorly to the sternal furcula; on a flat surface in the posterior and medial part of the acromion process; and one fixed at the junction of the deltoids attached with velcro to the volunteers' arm directly above the epicondyles of the humerus. A sensor will be connected to a stylus, for digitizing the anatomical points and constructing the coordinate system for each joint. The anatomical coordinate systems will be established for each segment by the digitization of the anatomical marks according to the protocol recommended by the International Society of Biomechanics - ISB36. The anatomical marks will be palpated and marked by a researcher who has experience with the protocol. then it will be estimated by passively moving the arm in short rotation amplitudes in several different positions. After completing the scan, the volunteers will assume a neutral standing position, with their arms resting in the body sludge, for approximately five seconds (time required for the angular values to be recorded).

The kinematic evaluation will be performed concomitantly with the recording of electromyographic activity. After the evaluation the subjects will be randomly distributed in Exercise Group (EG) and Biofeedback Group (BG) through the site www.randomization.com. GE and GB should attend twice a week, for eight consecutive weeks to the physiotherapy department of UFRN to carry out their respective intervention protocols. Each session will have an average duration of 30 minutes and should be justified in case of absence. All will be instructed to perform ice packs for 30 minutes in case of severe pain. The GE will perform a strengthening protocol and will have four elastic bands with different resistances available (light (red), moderate (blue), strong (purple) and extra strong (gray) for the progression of elbow flexion exercises, medial rotation of the shoulder, lateral rotation of the shoulder and scapular retraction. To determine the initial load the individual will perform a series of 10 repetitions of each exercise with the moderate resistance band (blue) and should not present pain greater than that reported in the initial evaluation and score above "moderate". For the exercise called "push up plus "the initial load will be determined from the kneeling position supported with the hands in the step using the same criteria of pain and scores of the borg scale mentioned above. The intensity progression will be due to the complexity of the exercise. Biofeedback (GB) volunteers will perform the same GE exercises added to the sEMG biofeedback in the upper trapezius (UT), Middle Trapezius (MT), Lower Trapezius (LT), and Anterior Serratil (AS) muscles in real time displayed in a computer screen during exercises. In the Y-axis of the screen the EMG amplitude is displayed and in the X-axis the time domain Volunteers will be instructed to change their movement strategies in order to decrease TS activity and facilitate MT, LT, and AS activity during exercises by viewing the computer screen. The researcher should guide the process through the verbal command.

ELIGIBILITY:
Inclusion Criteria:

* Present subacromial pain with a score greater than or equal to 2 (Visual Analog Scale) for more than 2 months;
* Positive Neer test;
* Positive Hawkins test;
* Positivie Jobe test (pain);
* Positive Patte test (pain);
* Involvement of the supraspinatus and / or infraspinatus tendon (without degenerative characteristics) confirmed by Magnetic Nuclear Resonance (MRI) examination.

Exclusion Criteria:

* Intense pain during the evaluations;
* Fail to properly perform the evaluation procedures;
* Two consecutive or five alternating absences during the training protocol.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Shouder pain | Change from baseline in shoulder pain at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluation of pain level in the shoulder using the Numerical Pain Scale, graded from 0 to 10, where 0 indicates absence of pain and 10 indicates the worst pain imaginable.
Shoulder function | Change from baseline in shoulder function at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluation of shoulder pain and function using the Disabilities of the Arm, Shoulder and Hand (DASH). The questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The higher the score, the greater the functional disability.

SECONDARY OUTCOMES:
Root Mean Square (RMS) | Change from baseline in RMS at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Analyze of the electromyographic activity of the shoulder complex muscles, after 4 and 8 weeks of the protocol and a follow up of 4 weeks after the intervention protocol, by Root Mean Square (RMS)
The kinematics of the scapula | Change from baseline in kinematics of the scapular girdle at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Analyze the kinematics of the scapula and glenohumeral in the slow and habitual movements after 4 and 8 weeks of the beginning of the protocol and a follow up of 4 weeks.
Peak of muscular torque | Change from baseline in peak of muscular torque at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluate the peak of muscular torque, after 4 and 8 weeks of the beginning of the protocol and a follow up of 4 weeks, using the hand-held dynamometer.
Peak torque time | Change from baseline in peak torque time at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Evaluate the peak torque time, after 4 and 8 weeks of the beginning of the protocol and a follow up of 4 weeks, using the hand-held dynamometer
Range of motion | Change from baseline in range of motion at 4 weeks, 8 weeks and follow up of 4 weeks after the intervention protocol
  Measure the range of motion for flexion, hyperextension, internal and external shoulder rotation after 4 and 8 weeks of the beginning of the protocol and a follow up of 4 weeks, using the inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Araken Oliveira, Ms, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (2):
- Brazil (2):
  - Jamilson Simões Brasileiro, Natal, Rio Grande do Norte
  - Araken kleber Azevedo de Oliveira, Parnamirim, Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No